CLINICAL TRIAL: NCT05395260
Title: A Pilot Window of Opportunity Trial: FL-101 in Non-Metastatic Muscle Invasive Bladder Cancer
Brief Title: FL- 101 Study in Non-Metastatic MIBC
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Flame Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-101-1003
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Muscle Invasive Bladder Carcinoma
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FL-101-IV (Experimental): Open Label Infusion of FL-101 on Day 1 and Day 15
  Interventions: Drug: FL-101

INTERVENTIONS:
Drug: FL-101 — FL-101 200mg IV

SUMMARY:
A pilot window of opportunity study of FL-101 in patients with non-metastatic MIBC who are eligible for radical cystectomy (RC) but are ineligible for, or decline, cisplatin-based neoadjuvant therapy.

DETAILED DESCRIPTION:
This is a pilot window of opportunity study of FL-101 in patients with non-metastatic MIBC who are eligible for radical cystectomy (RC) but are ineligible for, or decline, cisplatin-based neoadjuvant therapy.

The target recruitment will be 5 evaluable patients, with a possible expansion. Eligible patients will be enrolled to receive two doses of FL-101 prior to RC. FL-101 will be administered intravenously (IV) every two weeks (i.e., on Day 1 and Day 15).

Safety will be assessed by monitoring and recording all TEAEs graded by the NCI CTCAE v.5.0. In addition, laboratory assessments (hematology, serum chemistry, coagulation, and urinalysis), vital signs, physical exams, and 12-lead electrocardiogram (ECG) findings will be used to evaluate the safety of FL-101.

The PK of FL-101 will be characterized by analyzing samples collected at the time points.

To assess the immunogenicity of FL-101, ADAs will be measured as indicated in the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age.
* Able and willing to comply with protocol-specified requirements and to provide written informed consent.
* Patients must have histologically confirmed muscle-invasive bladder cancer (MIBC; T2-T4a, N0, M0 per American Joint Commission on Cancer [AJCC]) pure or mixed histology urothelial carcinoma [urothelial carcinoma should be the dominant histology].
* The initial TURBT that showed muscularis propria invasion should be within 12 weeks prior to beginning study therapy.
* Patients must have sufficient baseline tumor tissue from either initial or repeat TURBTs for submission of at least 20 unstained slides for translational study objectives. Patients with available unstained slides <20 may be considered on a case-by-case basis after discussion with the Sponsor (Note: An FFPE tissue block(s) may also be acceptable.
* Patients must be ineligible for cisplatin-based chemotherapy.
* Patients must be a candidate for radical cystectomy (RC) and planned to undergo RC per their treating physician
* C-reactive protein (CRP) level ≥5 mg/L
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function.
* Fully vaccinated against COVID-19 at least 4 weeks before the start of Screening activities. If under consideration for a booster, the booster administration needs to be complete within the same time constraint (ie, at least 4 weeks before the start of Screening activities).
* Adequate contraception for Men and Women or practice abstinence as well as refrain from donating sperm during the treatment period and for at least 180 days after the last dose of study treatment.
* Women may participate if not pregnant or breastfeeding.

Exclusion Criteria:

* Prior systemic therapy for muscle invasive UCB/MIBC
* Prior radiation therapy for muscle invasive UCB/MIBC
* Intravesical therapy within 6 weeks of Day 1 of trial
* Malignancies other than MIBC/muscle invasive UCB within 2 years prior to Day 1 of this trial, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate specific antigen [PSA] ≤ 10 mg/mL, etc.)
* Currently participating in or has participated in a trial of an investigational agent within 4 weeks prior to the first dose of study treatment or 5 half-lives, whichever is longer without recovery of clinically significant toxicities from that therapy.
* Known severe hypersensitivity (CTCAE v5.0, Grade ≥3) to FL-101, its active substance, or any of its excipients.
* Known history of human immunodeficiency virus or active Hepatitis B or Hepatitis C infection.
* Symptomatic herpes zoster within the past 30 days, a serious bacterial infection within the past 6 months or have had other recent or ongoing signs of infections.
* Received a live or attenuated vaccine within 30 days prior to the first dose of study treatment.
* Clinically unstable disease in any organ system despite current therapy, including, but not limited to ongoing or active infection including tuberculosis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations.
* Use of illicit drugs or excess intake of alcohol, based on the judgement of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Effect of FL-101 on CRP | Screening visit through 4 weeks post surgery day
  Evaluate the post-treatment changes in CRP from baseline

SECONDARY OUTCOMES:
The incidence of treatment emergent adverse events | Day 1 through up to 6 weeks post surgery day
  Safety and tolerability will be evaluated by incidence rate of treatment emergent adverse events of baseline.
Episodes of serious adverse events in patients with MIBC treated with FL-101 | Day 1 through up to 6 weeks post surgery day
  Safety and tolerability will be evaluated by the severity of treatment emergent adverse events of baseline.
Evaluate the concentration of FL-101 in whole blood | Day 1 through up to 6 weeks post surgery day
  Measure of concentration of FL-101 in whole blood at specific timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sumanta Kumar Pal, MD, Principal Investigator — City of Hope Comprehensive Center

IPD SHARING:
Plan to Share IPD: No